CLINICAL TRIAL: NCT06212999
Title: A Phase 3, Double-Blind Study to Evaluate the Long-Term Safety and Efficacy of Povorcitinib in Participants With Moderate to Severe Hidradenitis Suppurativa
Brief Title: A Study to Evaluate the Long-Term Safety and Efficacy of Povorcitinib in Participants With Moderate to Severe Hidradenitis Suppurativa
Acronym: STOP-HS LTE
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INCB 54707-312; 2023-507204-31-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2024-01-09; First posted 2024-01-19 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Hidradenitis Suppurativa (HS)
Keywords: Hidradenitis Suppurativa; Hidradenitis; Acne inversa; HS; Povorcitinib; Long-Term Extension (LTE); INCB054707
MeSH Terms: conditions — Hidradenitis Suppurativa; Hidradenitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Cohort C is open-label.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort A (Experimental): Povorcitinib at the protocol-defined dose strength based on cohort assignment.
  Interventions: Drug: Povorcitinib
- Cohort B (Experimental): Povorcitinib at the protocol-defined dose strength based on cohort assignment.
  Interventions: Drug: Povorcitinib
- Cohort C (Experimental): Povorcitinib at the protocol-defined dose strength based on cohort assignment.
  Interventions: Drug: Povorcitinib

INTERVENTIONS:
Drug: Povorcitinib — Oral; Tablet
  Other Names: INCB054707

SUMMARY:
The purpose of this study is to evaluate long-term safety and efficacy of povorcitinib in participants with moderate to severe hidradenitis suppurativa who completed the 54 weeks of study treatment within the originating parent Phase 3 studies (INCB 54707-301 [NCT05620823] or INCB 54707-302 [NCT05620836]).

ELIGIBILITY:
Inclusion Criteria:

* Completion of the study treatment period of the originating parent study (INCB 54707-301 or INCB 54707-302).
* Agreement to use contraception.
* Willing and able to comply with the study protocol and procedures.
* Further inclusion criteria apply.

Exclusion Criteria:

* Participation in the extension study could expose the participant to an undue safety risk.
* Women who are pregnant (or who are considering pregnancy) or breastfeeding.
* Further exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 617 (Actual)
Dates: Start 2024-01-30 (Actual); Primary Completion 2026-12-26 (Estimated); Study Completion 2026-12-26 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with Treatment-Emergent Adverse Events (TEAEs) | up to approximately 56 weeks
  TEAE is defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not it is considered drug-related. An AE can therefore be any unfavorable or unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study drug.

SECONDARY OUTCOMES:
Proportion of participants with Serious Treatment-Emergent Adverse Events (TEAEs) | up to approximately 56 weeks
  Serious TEAE is defined as any untoward medical occurrence that, at any dose, meet at least one of the following criteria: (a) results in death; (b) is life-threatening; (c) requires inpatient hospitalization or prolongation of existing hospitalization; (d) results in persistent or significant disability/incapacity; (e) is a congenital anomaly/birth defect; (f) is an important medical event.
Proportion of participants with TEAEs leading to study drug discontinuation | up to approximately 56 weeks
  Defined as any TEAE that leads to discontinuation of study drug.
Proportion of participants who achieve Hidradenitis Suppurativa Clinical Response (HiSCR) | up to approximately 56 weeks
  HiSCR is defined as at least a 50% reduction from baseline of parent study in the total abscess and inflammatory nodule (AN) count, with no increase from baseline of parent study in abscess or draining tunnel count.
Proportion of participants who achieve Hidradenitis Suppurativa Clinical Response 75 (HiSCR75) | up to approximately 56 weeks
  HiSCR75 is defined as at least a 75% reduction from baseline of parent study in the total AN count, with no increase from baseline of parent study in abscess or draining tunnel count.
Proportion of participants who achieve Hidradenitis Suppurativa Clinical Response 90 (HiSCR90) | up to approximately 56 weeks
  HiSCR90 is defined as at least a 90% reduction from baseline of parent study in the total AN count, with no increase from baseline of parent study in abscess or draining tunnel count.
Proportion of participants who achieve Hidradenitis Suppurativa Clinical Response 100 (HiSCR100) | up to approximately 56 weeks
  HiSCR100 is defined as a 100% reduction from baseline of parent study in the total AN count, with no increase from baseline of parent study in abscess or draining tunnel count.
Proportion of participants with flare at each visit | up to approximately 56 weeks
  Flare is defined as at least a 25% increase in the total AN count with a minimum increase of 2 ANs relative to Week 54.
Time to first flare | up to approximately 56 weeks
  Time to first flare during the long-term extension study.
Mean change from baseline of parent study in Hidradenitis Suppurativa Quality of Life (HiSQoL) score at each visit | up to approximately 56 weeks
  The HiSQoL is a HS-specific, health-related quality of life (QoL) instrument. The HiSQoL total score ranges from 0 to 68, with higher scores indicating higher disease impact on QoL.
Mean change from baseline of parent study in Dermatology Life Quality Index (DLQI) score at each visit | up to approximately 56 weeks
  The DLQI is a skin disease specific questionnaire aimed at the evaluation of how symptoms and treatment affect participants' health-related quality of life (QoL). The DLQI total score ranges from 0 to 30, with higher scores indicating lower skin health related QoL.
Proportion of participants with no increase in abscess and inflammatory nodule (AN) count relative to Week 54 at each visit | up to approximately 56 weeks
Proportion of participants with no increase in abscess, inflammatory nodule, and draining tunnel (ANdT) count relative to Week 54 at each visit | up to approximately 56 weeks
  ANdT count is defined as the total sum of abscesses, inflammatory nodules, and draining tunnels.
Proportion of participants with no increase in draining tunnel count relative to Week 54 at each visit | up to approximately 56 weeks
Proportion of participants with a total AN count of 0, 1, or 2 at each visit | up to approximately 56 weeks
  AN count defined as the total sum of abscesses and inflammatory nodules.
Proportion of participants with a total ANdT count of 0, 1, or 2 at each visit | up to approximately 56 weeks
  ANdT count is defined as the total sum of abscesses, inflammatory nodules, and draining tunnels.

CONTACTS AND LOCATIONS:
Overall Officials: Incyte Medical Monitor, Study Director — Incyte Corporation
Locations (165):
- United States (61):
  - Investigative Site US303, Phoenix, Arizona
  - Investigative Site US240, Scottsdale, Arizona
  - Investigative Site US307, Fort Smith, Arkansas
  - Investigative Site US214, Rogers, Arkansas
  - Investigative Site US315, Laguna Niguel, California
  - Investigative Site US223, Los Angeles, California
  - Investigative Site US222, Oakland, California
  - Investigative Site US226, San Diego, California
  - Investigative Site US309, Clearwater, Florida
  - Investigative Site US317, Hialeah, Florida
  - Investigative Site US306, Hollywood, Florida
  - Investigative Site US320, Hollywood, Florida
  - Investigative Site US316, Maitland, Florida
  - Investigative Site US227, Margate, Florida
  - Investigative Site US204, Miami, Florida
  - Investigative Site US236, Miami, Florida
  - Investigative Site US321, North Miami Beach, Florida
  - Investigative Site US200, Ocala, Florida
  - Investigative Site US228, Tampa, Florida
  - Investigative Site US201, Tampa, Florida
  - Investigative Site US311, Marietta, Georgia
  - Investigative Site US220, West Dundee, Illinois
  - Investigative Site US206, Indianapolis, Indiana
  - Investigative Site US337, Indianapolis, Indiana
  - Investigative Site US341, Bowling Green, Kentucky
  - Investigative Site US209, Louisville, Kentucky
  - Investigative Site US305, Baton Rouge, Louisiana
  - Investigative Site US207, Metairie, Louisiana
  - Investigative Site US229, New Orleans, Louisiana
  - Investigative Site US224, Baltimore, Maryland
  - Investigative Site US325, Marriottsville, Maryland
  - Investigative Site US225, Boston, Massachusetts
  - Investigative Site US304, Boston, Massachusetts
  - Investigative Site US310, Brighton, Massachusetts
  - Investigative Site US221, Quincy, Massachusetts
  - Investigative Site US213, Fort Gratiot, Michigan
  - Investigative Site US217, Waterford, Michigan
  - Investigative Site US212, Minneapolis, Minnesota
  - Investigative Site US302, St Louis, Missouri
  - Investigative Site US318, Portsmouth, New Hampshire
  - Investigative Site US230, East Windsor, New Jersey
  - Investigative Site US324, Kew Gardens, New York
  - Investigative Site US202, New York, New York
  - Investigative Site US210, Rochester, New York
  - Investigative Site US205, Chapel Hill, North Carolina
  - Investigative Site US215, Bexley, Ohio
  - Investigative Site US339, Bexley, Ohio
  - Investigative Site US330, Boardman, Ohio
  - Investigative Site US314, Cincinnati, Ohio
  - Investigative Site US312, Cleveland, Ohio
  - Investigative Site US203, Gahanna, Ohio
  - Investigative Site US301, Portland, Oregon
  - Investigative Site US232, Murfreesboro, Tennessee
  - Investigative Site US235, Arlington, Texas
  - Investigative Site US218, Bellaire, Texas
  - Investigative Site US340, Bellaire, Texas
  - Investigative Site US238, Pflugerville, Texas
  - Investigative Site US300, Plano, Texas
  - Investigative Site US234, San Antonio, Texas
  - Investigative Site US313, Norfolk, Virginia
  - Investigative Site US308, Spokane, Washington
- Australia (7):
  - Investigative Site AU203, Charlestown, New South Wales
  - Investigative Site AU205, Kogarah, New South Wales
  - Investigative Site AU200, Liverpool, New South Wales
  - Investigative Site AU206, Woolloongabba, Queensland
  - Investigative Site AU207, Woolloongabba, Queensland
  - Investigative Site AU201, Carlton, Victoria
  - Investigative Site AU204, Melbourne, Victoria
- Austria (2):
  - Investigative Site AT306, Inssbruck
  - Investigative Site AT305, Vienna
- Belgium (3):
  - Investigative Site BE300, Brussels
  - Investigative Site BE301, Ghent
  - Investigative Site BE302, Liège
- Bulgaria (5):
  - Investigative Site BG203, Sofia
  - Investigative Site BG202, Sofia
  - Investigative Site BG200, Sofia
  - Investigative Site BG204, Sofia
  - Investigative Site BG201, Stara Zagora
- Canada (14):
  - Investigative Site CA202, Calgary, Alberta
  - Investigative Site CA204, Edmonton, Alberta
  - Investigative Site CA200, Surrey, British Columbia
  - Investigative Site CA301, Winnipeg, Manitoba
  - Investigative Site CA205, Fredericton, New Brunswick
  - Investigative Site CA304, Barrie, Ontario
  - Investigative Site CA308, Hamilton, Ontario
  - Investigative Site CA303, London, Ontario
  - Investigative Site CA207, Mississauga, Ontario
  - Investigative Site CA302, Peterborough, Ontario
  - Investigative Site CA208, Richmond Hill, Ontario
  - Investigative Site CA307, Montreal, Quebec
  - Investigative Site CA206, Saint-Jérôme, Quebec
  - Investigative Site CA203, St. John's
- Czechia (2):
  - Investigative Site CZ301, Ostrava - Poruba
  - Investigative Site CZ300, Prague
- Denmark (2):
  - Investigative Site DK200, Århus N
  - Investigative Site DK201, Roskilde
- France (13):
  - Investigative Site FR305, Bordeaux
  - Investigative Site FR303, Brest
  - Investigative Site FR205, Dijon
  - Investigative Site FR307, Le Mans
  - Investigative Site FR204, Lyon
  - Investigative Site FR304, Marseille
  - Investigative Site FR302, Nantes
  - Investigative Site FR203, Nice
  - Investigative Site FR300, Paris
  - Investigative Site FR206, Reims
  - Investigative Site FR202, Rouen
  - Investigative Site FR301, Saint-Priest-en-Jarez
  - Investigative Site FR306, Toulouse
- Germany (15):
  - Investigative Site DE202, Berlin
  - Investigative Site DE203, Bochum
  - Investigative Site DE305, Darmstadt
  - Investigative Site DE201, Dessau
  - Investigative Site DE302, Dresden
  - Investigative Site DE306, Düsseldorf
  - Investigative Site DE207, Erlangen
  - Investigative Site DE301, Frankfurt
  - Investigative Site DE208, Göttingen
  - Investigative Site DE303, Hamburg
  - Investigative Site DE300, Hanover
  - Investigative Site DE205, Heidelberg
  - Investigative Site DE200, Kiel
  - Investigative Site DE307, Memmingen
  - Investigative Site DE206, Merzig
- Greece (3):
  - Investigative Site GR300, Athens
  - Investigative Site GR303, Athens
  - Investigative Site GR302, Thessaloniki
- Italy (6):
  - Investigative Site IT200, Ancona
  - Investigative Site IT207, Catania
  - Investigative Site IT202, Milan
  - Investigative Site IT206, Pisa
  - Investigative Site IT205, Roma
  - Investigative Site IT201, Rozzano
- Japan (8):
  - Investigative Site JP301, Ginowan-shi
  - Investigative Site JP304, Itabashi-ku
  - Investigative Site JP305, Kurume-shi
  - Investigative Site JP300, Kyoto
  - Investigative Site JP303, Niigata
  - Investigative Site JP308, Sapporo
  - Investigative Site JP302, Sendai
  - Investigative Site JP309, Shinjuku-ku
- Netherlands (3):
  - Investigative Site NL302, Breda
  - Investigative Site NL303, Groningen
  - Investigative Site NL301, Rotterdam
- Poland (7):
  - Investigative Site PL203, Lublin
  - Investigative Site PL304, Ostrowiec Świętokrzyski
  - Investigative Site PL200, Rzeszów
  - Investigative Site PL201, Warsaw
  - Investigative Site PL202, Warsaw
  - Investigative Site PL301, Wroclaw
  - Investigative Site PL302, Wroclaw
- Spain (11):
  - Investigative Site ES203, Alicante
  - Investigative Site ES302, Badalona
  - Investigative Site ES303, Barcelona
  - Investigative Site ES301, Granada
  - Investigative Site ES202, Las Palmas de Gran Canaria
  - Investigative Site ES201, Madrid
  - Investigative Site ES205, Madrid
  - Investigative Site ES305, Madrid
  - Investigative Site ES200, Manises
  - Investigative Site ES300, Pontevedra
  - Investigative Site ES304, Santiago de Compostela
- United Kingdom (3):
  - Investigative Site GB202, Birmingham
  - Investigative Site GB200, Dudley
  - Investigative Site GB203, Salford

IPD SHARING:
Plan to Share IPD: Yes
Incyte shares data with qualified external researchers after a research proposal is submitted. These requests are reviewed and approved by a review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  The trial data availability is according to the criteria and process described on https://www.incyte.com/our-company/compliance-and-transparency
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the primary publication or 2 years after the study has ended for market authorized products and indications.
Access Criteria: Data from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.incyteclinicaltrials.com website. For approved requests, the researchers will be granted access to anonymized data under the terms of a data sharing agreement.
URL: https://www.incyte.com/our-company/compliance-and-transparency

REFERENCES:
- See also: A Study to Evaluate the Long-Term Safety and Efficacy of Povorcitinib in Participants With Moderate to Severe Hidradenitis Suppurativa (STOP-HS LTE) — https://www.incyteclinicaltrials.com/study/?id=INCB%2054707-312&SearchTerm=INCB%2054707-312&Latitude=&Longitude=&LocationName=&conditions=&Status=&phases=&AgeRanges=&gender=&StudyTypes=&AttachmentTypes=&MileRadius=100&PageIndex=0&PageSize=10&SortField=&SortOrder=&hasResults=